CLINICAL TRIAL: NCT07164716
Title: Immediate Myofascial Responses to Plantar Fascia Recovery Training in Adolescent Endurance Runners: A Dorsal Chain Perspective
Brief Title: Immediate Myofascial Responses to PFRT in Adolescent Endurance Runners
Acronym: PFRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kübra Sarıoğlu, Sub-Investigator, Kübra Sarıoğlu, PT, MSc (PhD student), Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HU-FTR-KS-02
Record Dates: First submitted 2025-08-12; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Recovery, Psychological
Keywords: plantar fascia; fascial chain; bunkie test; superficial back muscles; myofascial release; running

STUDY DESIGN:
Intervention Model Description: There were two running groups: one received the treatment and was tested, while the other served as the control group.
Who Masked: Participant
Masking Description: A randomized controlled trial included 34 adolescent runners, with 17 in the plantar fascia recovery training (PFRT) group and 17 in the control group. After running training, the PFRT group received bilateral PFRT. Assessments were conducted pre-training, post-training, and post-PFRT on the dominant side. DKCP was evaluated using the Bunkie Test for the posterior power line (PPL) and posterior stabilization line (PSL), Myoton measurements for latissimus dorsi (LD), erector spinae, hamstrings, and gastrocnemius, the Sit-and-Reach Test for hamstring and lumbar flexibility, and the Modified Schober Test for lumbar mobility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plantar fascia recovery training group (Experimental): Foam roller, Metatarsophalangeal Joint Stretching, Soft tissue mobilization, Gliding massage
  Interventions: Other: plantar fascia recovery training group
- control group (No Intervention)

INTERVENTIONS:
Other: plantar fascia recovery training group — plantar fascia recovery training group: Gliding massage,Soft tissue mobilization,Metatarsophalangeal Joint Stretching,Foam roller
  Arms: plantar fascia recovery training group

SUMMARY:
This study aimed to investigate the acute effects of post-run plantar fascia recovery training (PFRT) on dorsal kinetic chain performance (DKCP) in adolescent long-distance runners. In the study, runners divided into two groups were assessed before training, after training, and following the plantar fascia intervention. The effects on both the performance and flexibility of the muscle and connective tissues of the back and posterior leg were examined.

DETAILED DESCRIPTION:
This study aimed to investigate the acute effects of post-run plantar fascia recovery training (PFRT) on dorsal kinetic chain performance (DKCP) in adolescent long-distance runners. A randomized controlled trial was conducted with 34 adolescent runners, divided equally into a PFRT group and a control group. Following running training, the PFRT group received bilateral PFRT. Assessments were performed pre-training, post-training, and post-PFRT on the dominant side. DKCP was evaluated using the Bunkie Test for the posterior power line (PPL) and posterior stabilization line (PSL), Myoton measurements for the latissimus dorsi, erector spinae, hamstrings, and gastrocnemius muscles, the Sit-and-Reach Test for hamstring and lumbar flexibility, and the Modified Schober Test for lumbar mobility.

ELIGIBILITY:
Inclusion Criteria:

* participating as a long-distance runner
* between 14 and 18 years old
* running a weekly distance between 30-60 km
* having at least 2 years of regular running training experience

Exclusion Criteria:

• having any chronic illness or a history of lower extremity and/or spinal injury in the past 6 months

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Bunkie Test | Pre-training, Post-training, Post-intervention. Pre-training: 30 minutes before training Post-training (Immediate): Immediately after training Post-intervention: 10 minutes after intervention
  Participants hold specific Bunkie Test positions engaging PPL(posterior power line) and PSL (posterior stabilization line )muscles. Maximum hold time is recorded for each position, up to a limit of 40 seconds.

SECONDARY OUTCOMES:
Muscle mechanical properties assessed using the MyotonPRO device. | Pre-training, Post-training, Post-intervention Pre-training: 30 minutes before training Post-training (Immediate): Immediately after training Post-intervention: 10 minutes after intervention
  The MyotonPRO handheld device provides quantitative measurements of muscle tone, stiffness, and elasticity at the target muscle sites. Measurements are taken according to standard protocols immediately before and after the intervention. Muscle mechanical properties, including tone (Hz), stiffness (N/m), and elasticity (unitless, measured as logarithmic decrement), were assessed using the MyotonPRO device

OTHER OUTCOMES:
Sit and Reach Test. | Pre-training, Post-training, Post-intervention Pre-training: 30 minutes before training Post-training (Immediate): Immediately after training Post-intervention: 10 minutes after intervention
  Hamstring and lower back flexibility assessed using the Sit and Reach Test. Participants perform the Sit and Reach Test following standard protocols. The maximum distance reached (in centimeters) is recorded. Three trials are conducted, and the best value is used for analysis.
Modified Schober Test | Pre-training, Post-training, Post-intervention Pre-training: 30 minutes before training Post-training (Immediate): Immediately after training Post-intervention: 10 minutes after intervention
  Lumbar spine flexion mobility assessed using the Modified Schober Test. Participants perform forward trunk flexion, and the change in distance (cm) between marked points on the lumbar spine is measured. Maximum flexion achieved during the test is recorded.
Demografic Information, age of participants | Baseline
  Age of participants, Mean age (years) of participants in PFRT and Control groups at baseline.
Height of participants | Baseline
  Mean height (meters) of participants in PFRT and Control groups at baseline.
Body weight of participants | Baseline
  Mean body weight (kilograms) of participants in PFRT and Control groups at baseline.
Body Mass Index (BMI) of participants | Baseline
  Mean BMI (kg/m²) of participants in PFRT and Control groups at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: KÜBRA SARIOĞLU, Msc, Principal Investigator — HACETTEPE ÜNİVERSİTESİ ,Anafartalar, Talatpaşa Blv No:47, 06100 Altındağ/Ankara
Locations (1):
- Hacettepe Üniversitesi Fizik Tedavi Ve Rehabilitasyon Fakültesi Sporcu Sağlığı Ünitesi, Ankara, ÇANKAYA, Turkey (Türkiye)